CLINICAL TRIAL: NCT01505101
Title: Mindfulness-Oriented Recovery Enhancement for Chronic Pain Patients Receiving Opioid Therapy: Exploration of Cognitive, Affective, and Physiological Mechanisms
Brief Title: Mindfulness-Oriented Recovery Enhancement for Chronic Pain Patients Receiving Opioid Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Fahs Beck Fund for Research and Experimentation (Unknown)
Responsible Party: Principal Investigator, Eric Garland, Assistant Professor, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DA032517-01; R03DA032517 (NIH)
Record Dates: First submitted 2012-01-04; First posted 2012-01-06 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-08

CONDITIONS: Chronic Pain; Opioid Abuse, Unspecified Use
MeSH Terms: conditions — Chronic Pain; Opioid-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mindfulness-Oriented Recovery Enhancement (Experimental)
  Interventions: Behavioral: Mindfulness-Oriented Recovery Enhancement
- Conventional Support Group (SG) (Active Comparator)
  Interventions: Behavioral: Conventional Support Group (SG)

INTERVENTIONS:
Behavioral: Mindfulness-Oriented Recovery Enhancement — MORE is a multimodal, dual-process group intervention involving mindfulness training, cognitive restructuring, and positive emotion induction. MORE consists of eight, weekly, two-hour group sessions led by a trained therapist.
  Arms: Mindfulness-Oriented Recovery Enhancement
Behavioral: Conventional Support Group (SG) — The control arm will participate in a time-matched, conventional SG led by a Master's level therapist, discussing topics pertinent to chronic pain and opioid misuse. The SG format is adapted from the support group detailed in the evidence-based, Matrix Intensive Outpatient Treatment manual. The SG consists of eight, weekly, two-hour sessions.
  Arms: Conventional Support Group (SG)

SUMMARY:
Persons suffering from chronic pain who are treated with long-term opioid therapy are at risk of misusing prescription opioids and developing opioid addiction. Moreover, long-term use of opioids may result in hyperalgesia, which exacerbates opioid craving and consumption. Mindfulness interventions have been shown reduce chronic pain symptoms, addictive processes, and substance use. The investigators hypothesize that relative to a support group control condition, participation in a novel mindfulness-oriented cognitive intervention, Mindfulness-Oriented Recovery Enhancement (MORE), will result in improved well-being and decreased pain, opioid craving, and opioid misuse behaviors among chronic pain patients receiving opioid therapy.

DETAILED DESCRIPTION:
Few behavioral treatments target the cognitive-affective mediators of opioid misuse and addiction in chronic pain patients. As such, novel, multimodal interventions are needed to effectively target key mechanisms in the risk chain from chronic pain to opioid misuse and addiction. The secondary aim of this study is to explore possible cognitive, affective, and psychophysiological mediators of intervention effects on pain, opioid craving, opioid misuse behaviors, and well-being.

ELIGIBILITY:
Inclusion Criteria:

* chronic pain diagnosis (ICD-9 diagnoses 338.xx)
* treatment with prescription opioids for > 3 months

Exclusion Criteria:

* prior mindfulness training
* persons who are experiencing acute opioid withdrawal
* suicidal ideation
* psychosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2011-10; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Pain severity, pain functional interference | Baseline, immediately following treatment, and at 3 month follow-up
  Change in pain severity, functional interference, and relief from pain treatments measured on the Brief Pain Inventory-Short Form.
Opioid craving | Baseline, immediately following treatment, and at 3 month follow-up
  Change in opioid craving as measured by the Obsessive-Compulsive Drug Use Scale and a single-item measure of instantaneous craving.
Opioid misuse behaviors | Baseline, immediately following treatment, and at 3 month follow-up
  Change in opioid misuse behaviors as measured by the Current Opioid Misuse Measure
Well-being | Baseline, immediately following treatment, and at 3 month follow-up
  Change in well-being as measured by the WHO-5

SECONDARY OUTCOMES:
Attentional bias | Baseline and immediately following treatment
  Change in attentional bias as measured by a dot probe task
Psychophysiological cue-reactivity | Baseline and immediately following treatment
  Change in psychophysiological cue-reactivity
Emotional response inhibition | Baseline and immediately following treatment
  Change in emotional response inhibition
Pain coping strategies | Baseline, intervention midpoint, and immediately following treatment
  Change in reinterpretation of pain sensations, catastrophizing, and suppression.
Anhedonia | Baseline and immediately following treatment
  Change in anhedonia
Fear of pain | Baseline and immediately following treatment
  Change in fear of pain
Mindfulness | Baseline, intervention midpoint, and immediately following treatment
  Change in mindfulness measured by the Five-Facet Mindfulness Questionnaire and the Toronto Mindfulness Scale
Positive reappraisal | Baseline and immediately following treatment
  Change in positive reappraisal

CONTACTS AND LOCATIONS:
Overall Officials: Eric L Garland, PhD, Principal Investigator — Florida State University
Locations (1):
- FSU College of Social Work, Tallahassee, Florida, United States